CLINICAL TRIAL: NCT01094561
Title: Secretin-Stimulated MRCP as an Early Screening Modality for Pancreatic Ductal Abnormalities in Patients at High Risk for Pancreatic Adenocarcinoma: A Pilot Study
Brief Title: Secretin-Stimulated Magnetic Resonance Cholangiopancreatography (S-MRCP) in Pancreatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Hecht (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Hecht, Associate Professor of Clinical Radiology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAC1038
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Results first posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: Family history of pancreatic cancer; Pancreatic adenocarcinoma; Imaging techniques; Synthetic human secretin; Pancreatic abnormalities; Early detection and prevention
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Synthetic Human Secretin (Experimental): Single arm (open label).
  Interventions: Drug: Synthetic Human Secretin; Procedure: Secretin-Enhanced Magnetic Resonance Cholangiopancreatography; Procedure: Secretin-Enhanced Endoscopic Ultrasound

INTERVENTIONS:
Drug: Synthetic Human Secretin — Subjects will each undergo a Secretin-Enhanced Magnetic Resonance Cholangiopancreatography (S-MRCP) and a Secretin-Enhanced Endoscopic Ultrasound (S-EUS) evaluation, at a dose of 0.2 ucg/kg per exam. Synthetic Human Secretin, provided by the Repligen Corporation, will be administered by IV bolus injection over 30 seconds followed by a 30 second saline flush. The maximum dose of secretin will be 18.5 ucg.
  Other Names: RG1068
Procedure: Secretin-Enhanced Magnetic Resonance Cholangiopancreatography
  Other Names: S-MRCP
Procedure: Secretin-Enhanced Endoscopic Ultrasound
  Other Names: S-EUS

SUMMARY:
The aim of our study is to evaluate the utility of Secretin-Stimulated Magnetic Resonance Cholangiopancreatography (S-MRCP) in detecting carcinoma and precancerous lesions in patients with a significant family history of pancreatic adenocarcinoma. Our hypothesis is that S-MRCP is superior to traditional computed tomography (CT) or magnetic resonance imaging (MRI) in detecting early pancreatic neoplasms, and approaches the accuracy of endoscopic ultrasound (EUS).

DETAILED DESCRIPTION:
Pancreatic cancer remains the fourth leading cause of cancer-related death in the United States, largely due to the lack of accurate and cost-effective screening methods. Initial screening efforts should be directed at patients with known increased genetic risk for pancreatic adenocarcinoma. About 10-20% of pancreatic cancers are considered familial or syndromic. Since pancreatic adenocarcinoma is known to progress from preneoplastic lesions, termed pancreatic intraepithelial neoplasia (PanIN), it may eventually be possible to identify and cure patients by detecting preneoplastic lesions. Traditional radiological methods lack the resolution to detect early lesions. The sensitivity and specificity of endoscopic retrograde cholangiopancreatography (ERCP) (92%,96%) and EUS (93-98%)are better, but these procedures are invasive and limited in availability. Magnetic resonance cholangiopancreatography (MRCP) has emerged as a widely-accepted alternative with comparable sensitivity to ERCP. Magnetic Resonance Cholangiopancreatography (MRCP) has been further augmented by secretin stimulation, which improves visualization of the pancreatic duct as well as side branches. We will recruit 25 patients for a prospective pilot study examining S-MRCP as a screening technique in high-risk individuals. All recruited patients will undergo S-MRCP in conjunction with magnetic resonance imaging (MRI)/magnetic resonance angiography (MRA), as well as secretin-enhanced EUS (S-EUS). Those patients with abnormalities on S-MRCP or S-EUS will undergo ERCP. If ERCP also shows abnormalities, these patients will be recommended total or subtotal pancreatectomy. The primary outcome that we will be studying will be concordance of S-MRCP and EUS. Secondarily, we will be measuring positive predictive value of S-MRCP, in comparison with EUS and ERCP in identifying neoplasm in those patients who undergo surgical resection during this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older.
* At least two first or two second degree relatives with pancreatic adenocarcinoma (the study subject will be either 10 years younger than the youngest age at which a relative was diagnosed with pancreatic cancer, or the study subject will be at least 25 years of age).
* Fulfills criteria or has undergone genetic testing which confirms BRCA1 (BReast CAncer gene 1), BRCA2 (BReast CAncer gene 2), Familial Atypical Multiple Mole Melanoma, PeutzJeghers, Hereditary nonpolyposis colorectal cancer (HNPCC), Hereditary Pancreatitis, or ataxiatelangiectasia.

Exclusion Criteria:

* Any contraindication to MRI, including but not limited to implanted metal devices (e.g. pacemaker,berry aneurysm clips, neural stimulator or cochlear implants).
* Known pancreatic malignancy or dysplasia.
* Pregnancy.
* History of sensitivity to secretin.
* Creatinine greater than 2.
* Unwillingness or inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-07; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hecht, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were accrued from June 2007 to April 2011. All subjects were accrued and followed at Columbia University Medical Center.
Groups:
- Synthetic Human Secretin: Single arm (open label).
  Subjects will each undergo an S-MRCP and an S-EUS evaluation, at a dose of 0.2 ucg/kg per exam. Synthetic Human Secretin, provided by the Repligen Corporation, will be administered by IV bolus injection over 30 seconds followed by a 30 second saline flush. The maximum dose of secretin will be 18.5 ucg.
Period: Overall Study
Arm/Group | Synthetic Human Secretin
Started | 23
Completed | 17
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Synthetic Human Secretin
Number analyzed (Participants) | 23
Age, Customized [Number; unit: participants]
  18-29 years | 0
  30-39 years | 1
  40-49 years | 2
  50-59 years | 9
  >60 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: S-MRCP and S-EUS Concordance
Description: The primary outcome studied will be the concordance of S-MRCP and S-EUS. Screening will consist of two diagnostic imaging modalities. First, all patients will have S-MRCP in conjunction with contrast-enhanced magnetic resonance imaging (MRI)/magnetic resonance angiography (MRA). All images will be analyzed by a radiologist. Within thirty days, all patients will also undergo EUS with and without secretin enhancement (S-EUS).If the S-EUS shows abnormalities, EUS-guided fine-needle aspiration will be performed. The S-MRCP and EUS image findings will be classified as benign or suspicious/malignant to determine the concordance between imaging techniques.
  Due to poor enrollment, inadequate data was collected for data analysis and therefore data analysis was not conducted. There is no data to report.
Time Frame: Day 1 and up to 30 days after S-MRCP
Groups:
- Synthetic Human Secretin: Single arm (open label).
  Synthetic Human Secretin: Twenty five patients will each undergo an S-MRCP and an S-EUS evaluation, at a dose of 0.2 ucg/kg per exam. Synthetic Human Secretin, provided by the Repligen Corporation, will be administered by IV bolus injection over 30 seconds followed by a 30 second saline flush. The maximum dose of secretin will be 18.5 ucg.
Arm/Group | Synthetic Human Secretin
Number analyzed (Participants) | 0

2. Secondary Outcome: The Positive Predictive Value of S-MRCP
Description: The secondary outcome endpoints of our study will be positive predictive value of S-MRCP, in comparison with EUS/S-EUS and endoscopic retrograde cholangiopancreatography (ERCP), utilizing surgical pathology as the gold standard. In addition, we will also be looking at the utility of Cancer Antigen 19-9 (CA 19-9) and oral glucose tolerance tests.
  Due to poor enrollment, inadequate data was collected for data analysis and therefore data analysis was not conducted. There is no data to report.
Time Frame: Up to 1 year
Arm/Group | Synthetic Human Secretin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Synthetic Human Secretin
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes